CLINICAL TRIAL: NCT00858819
Title: Clinical Trial of Osteoporosis in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: VGFOUREG11961
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Ankylosing Spondylitis
Keywords: Osteoporosis; Fractures; Bone Mineral Density; Quantitative Computed Tomography
MeSH Terms: conditions — Spondylitis, Ankylosing; Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AS: Patients with AS attending three different rheumatology clinics in Western Sweden have been invited to participate.

SUMMARY:
This is an observational study aiming to study the prevalence and risk factors for osteoporosis and vertebral fractures in patients with ankylosing spondylitis attending three Rheumatology clinics in Western Sweden.

DETAILED DESCRIPTION:
Background Ankylosing spondylitis (AS) is a common inflammatory rheumatic disease with a prevalence of 0.5-1.0%. Men are more commonly affected by the disease as compared to women, ratio 2.6-4:1. Pain in the back is a frequent symptom of debut. This pain is often associated with sacroilitis. In later stages also the lumbar, thoracic and cervical spine are hit by the disease. Peripheral joints, eyes, heart, lungs and urinary tract may also be influenced.

Osteoporosis in AS In AS the risk of osteoporosis is increased. However, this field has not yet been significantly studied probably due to several reasons such as the predominance of men with the disease and men are more seldom investigated for osteoporosis compared to women. When AS progresses syndesmophytes of the spine are developed which makes it difficult to assess bone mineral density (BMD) correctly with the conventional method, dual energy x-ray absorptiometry (DXA). Fractures in the spine are easy to foreseen since the pain of the patient might be misjudged to be related to increased disease activity. Fractures are also overlooked in radiographs in AS. AS is associated with both increased bone formation and increased bone resorption. The bone remodeling process in the spine renders the spine less flexible and stiffer and as a consequence also a quite small trauma may result in a fracture. These fractures are often instable risking injuring the spinal cord and nerves.

Aims of the study

* To investigate the prevalence of osteoporosis and osteoporosis related fractures in patients with AS in Western Sweden.
* To identify risk factors for osteoporosis and osteoporosis related fractures in AS.
* To study how fractures in the spine may influence the pain in the back, the flexibility of the spine and the posture of the patients.
* To study to which extent the patients with AS are investigated and treated for osteoporosis.
* To investigate which method is most reliable for measuring BMD in AS.

Design and methods This is an observational study consisting of questionnaires, examination of the patients, blood tests, measures of BMD with different techniques, DXA, both frontal-dorsal and lateral projections, Quantitative Computed Tomography (QCT) and Xtreme CT. Patients with AS from three rheumatology clinics in western Sweden with definite AS will be invited to participate. It is estimated that about 250 patients will be included in the trial. All patients gave informed written consent according to the Declaration of Helsinki. The study has been approved by the Regional Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Definitive Ankylosing spondylitis according to the New York criteria
* At least 18 years old

Exclusion Criteria:

* Pregnant
* Dementia
* Not able to understand, speak or read Swedish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with definitive ankylosing spondylitis attending three rheumatology clinics in Western Sweden.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The prevalence of osteoporosis and osteoporosis related fractures in patients with AS in Western Sweden. | October 2009

SECONDARY OUTCOMES:
To investigate which method is the most reliable for measuring bone mineral density in ankylosing spondylitis | May 2010

CONTACTS AND LOCATIONS:
Overall Officials: Helena Forsblad d'Elia, Md, PhD, Principal Investigator — Department of Rheumatology and Inflammation Research
Locations (1):
- Department of Rheumatology and Inflammation Research, Gothenburg, Sweden

REFERENCES:
- [Derived] Klingberg E, Magnusson MK, Strid H, Deminger A, Stahl A, Sundin J, Simren M, Carlsten H, Ohman L, Forsblad-d'Elia H. A distinct gut microbiota composition in patients with ankylosing spondylitis is associated with increased levels of fecal calprotectin. Arthritis Res Ther. 2019 Nov 27;21(1):248. doi: 10.1186/s13075-019-2018-4. PMID 31771630
- [Derived] Law L, Beckman Rehnman J, Deminger A, Klingberg E, Jacobsson LTH, Forsblad-d'Elia H. Factors related to health-related quality of life in ankylosing spondylitis, overall and stratified by sex. Arthritis Res Ther. 2018 Dec 27;20(1):284. doi: 10.1186/s13075-018-1784-8. PMID 30587228
- [Derived] Torres L, Klingberg E, Nurkkala M, Carlsten H, Forsblad-d'Elia H. Hepatocyte growth factor is a potential biomarker for osteoproliferation and osteoporosis in ankylosing spondylitis. Osteoporos Int. 2019 Feb;30(2):441-449. doi: 10.1007/s00198-018-4721-4. Epub 2018 Oct 10. PMID 30306221
- [Derived] Deminger A, Klingberg E, Geijer M, Gothlin J, Hedberg M, Rehnberg E, Carlsten H, Jacobsson LT, Forsblad-d'Elia H. A five-year prospective study of spinal radiographic progression and its predictors in men and women with ankylosing spondylitis. Arthritis Res Ther. 2018 Aug 3;20(1):162. doi: 10.1186/s13075-018-1665-1. PMID 30075808
- [Derived] Klingberg E, Strid H, Stahl A, Deminger A, Carlsten H, Ohman L, Forsblad-d'Elia H. A longitudinal study of fecal calprotectin and the development of inflammatory bowel disease in ankylosing spondylitis. Arthritis Res Ther. 2017 Feb 2;19(1):21. doi: 10.1186/s13075-017-1223-2. PMID 28148281